CLINICAL TRIAL: NCT00006368
Title: A Phase I, Open-Label, Maximum Tolerated Single-Cycle and Four-Cycle Dose-Finding Study to Evaluation the Safety and Tolerability of 90Y-SMT 487 Administered by Intravenous Infusion to Subjects With Refractory Somatostatin-Receptor Positive Tumors
Brief Title: Yttrium Y 90 SMT 487 in Treating Patients With Refractory or Recurrent Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Purpose: Treatment
Other Study IDs: NOVARTIS-SMT-B151; MCC-12275; MCC-IRB-5473; CDR0000068241 (Registry Identifier: PDQ (Physician Data Query)); NCI-G00-1857
Record Dates: First submitted 2000-10-04; First posted 2004-04-02 (Estimated); Last update posted 2013-05-01 (Estimated); Status verified 2013-04

CONDITIONS: Brain and Central Nervous System Tumors; Breast Cancer; Gastrointestinal Carcinoid Tumor; Islet Cell Tumor; Lung Cancer; Lymphoma; Melanoma (Skin); Neoplastic Syndrome
Keywords: stage IV adult Hodgkin lymphoma; stage IV breast cancer; recurrent breast cancer; recurrent non-small cell lung cancer; recurrent adult Hodgkin lymphoma; extensive stage small cell lung cancer; recurrent small cell lung cancer; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; gastrinoma; recurrent adult brain tumor; insulinoma; recurrent islet cell carcinoma; ACTH-producing pituitary tumor; prolactin-producing pituitary tumor; growth hormone-producing pituitary tumor; recurrent pituitary tumor; TSH producing pituitary tumor; nonfunctioning pituitary tumor; adult brain stem glioma; adult craniopharyngioma; adult medulloblastoma; adult meningioma; adult glioblastoma; stage IV melanoma; recurrent melanoma; stage IV non-small cell lung cancer; WDHA syndrome; somatostatinoma; pancreatic polypeptide tumor; glucagonoma; pulmonary carcinoid tumor; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; adult anaplastic astrocytoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult central nervous system germ cell tumor; adult pilocytic astrocytoma; adult subependymoma; adult ependymoblastoma; adult pineocytoma; adult pineoblastoma; adult meningeal hemangiopericytoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; adult choroid plexus tumor; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult grade III meningioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Breast Neoplasms; Adenoma, Islet Cell; Lung Neoplasms; Lymphoma; Melanoma; Neoplasms; Hodgkin Disease; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Gastrinoma; Brain Neoplasms; Insulinoma; Carcinoma, Islet Cell; Growth Hormone-Secreting Pituitary Adenoma; Pituitary Neoplasms; Craniopharyngioma; Medulloblastoma; Meningioma; Glioblastoma; Vipoma; Somatostatinoma; Glucagonoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma, Subependymal; Neuroectodermal Tumors, Primitive; Pinealoma; Lymphoma, Mantle-Cell; Choroid Plexus Neoplasms; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Gliosarcoma | interventions — 90Y-octreotide, DOTA-Tyr(3)-

INTERVENTIONS:
Radiation: yttrium Y 90-edotreotide

SUMMARY:
RATIONALE: Radiolabeled drugs such as yttrium Y 90 SMT 487 can locate tumor cells and deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of yttrium Y 90 SMT 487 in treating patients who have refractory or recurrent cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of yttrium Y 90-SMT 487 in patients with recurrent malignant neoplasms that prove positive for somatostatin receptors. II. Determine the safety and lifetime serious adverse event profile of this regimen in these patients. II. Determine the antitumor effect and the effect of repeated administrations on the renal excretion pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose escalation, multicenter study. Patients undergo octreotide scintigraphy to determine the location of somatostatin receptors. Patients then receive yttrium Y 90-SMT 487 IV over 15 minutes on day 1. Treatment continues every 6 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients each are entered on course I (vertical dose escalation) and courses II, III, and IV (horizontal dose escalation). Cohorts receive escalating doses of yttrium Y 90-SMT 487 until the maximum tolerated dose (MTD) is determined. MTDs are determined for a single course and for 4 courses. The MTD is defined as the dose preceding that at which no more than 2 of 6 patients experience dose limiting toxicities. Results of course I determine the dosage of subsequent courses. Patients are evaluated on days 2 and 7, and at weeks 4 and 6, following each injection of yttrium Y 90-SMT 487. Patients are followed at 12 and 18 months and then annually thereafter.

PROJECTED ACCRUAL: Approximately 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed, progressive malignant neoplasm Clinical diagnosis of multiple endocrine neoplasia (MEN) types I and II allowed Tumors positive for somatostatin receptors by octreotide scintigraphy, such as: Pituitary Brain Endocrine pancreatic Lymphoma Carcinoid Melanoma Small cell lung Breast Disease not amenable to standard treatment OR Failed existing first and second line therapies (failed at least 1 regimen in the case of small cell lung cancer) Bone disease (no diffuse bone marrow involvement), pleural effusions, and ascites allowed

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Course I: Karnofsky 50-100% Courses II-IV: Karnofsky 30-100% Life expectancy: At least 6 months and no greater than 2.5 years (for course I only) Hematopoietic: Course I: Hemoglobin at least 8 g/dL WBC at least 3,500/mm3 Platelet count at least 100,000/mm3 Courses II-IV: WBC at least 3,000/mm3 Platelet count at least 75,000/mm3 Hepatic: Not specified Renal: Creatinine no greater than 1.7 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No history of congestive heart failure unless ejection fraction at least 40% Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for 6 months after study No other concurrent malignancy except MEN I or II or squamous cell skin cancer No concurrent significant, uncontrolled, medical, psychiatric, or surgical condition that would preclude study (course 1)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy Greater than 4 weeks since prior chemotherapy Endocrine therapy: At least 4 months since prior long acting somatostatin analogue Concurrent hormonal therapy (except somatostatin analogues) allowed if started at least 2 months previously Radiotherapy: Greater than 4 weeks since prior radiotherapy No prior radiotherapy to at least 25% of bone marrow Surgery: Greater than 4 weeks since prior surgery Other: Greater than 4 weeks since prior investigational drugs No other concurrent investigational drug therapy No other concurrent antineoplastic therapy Concurrent bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 1998-01; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry K. Kvols, MD, Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States